CLINICAL TRIAL: NCT01271816
Title: Prolonged Monitoring to Detect Ventricular Arrhythmias in Presymptomatic ARVC Patients
Brief Title: Prolonged Monitoring to Detect Ventricular Arrhythmias in Presymptomatic Arrhythmogenic Right Ventricular Cardiomyopathy (ARVC) Patients
Acronym: PREPARE
Status: Terminated | Type: Observational
Why Stopped: inadequate recruitment
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Collaborators: Abbott Medical Devices (Industry)
Responsible Party: Principal Investigator, Andrew Krahn, principal investigator, London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's
Other Study IDs: R-10-532; 17390 (Other: REB)
Record Dates: First submitted 2011-01-04; First posted 2011-01-07 (Estimated); Last update posted 2014-01-03 (Estimated); Status verified 2014-01

CONDITIONS: Arrhythmogenic Right Ventricular Cardiomyopathy (ARVC)
Keywords: genetics; sudden death; monitoring; loop recorder; cardiomyopathy
MeSH Terms: conditions — Arrhythmogenic Right Ventricular Dysplasia; Death, Sudden; Cardiomyopathies

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Presymptomatic ARVC gene carriers: ARVC gene positive patients without manifest ARVC after standard screening clinical testing.

SUMMARY:
Arrhythmogenic Right Ventricular Cardiomyopathy (ARVC) is an inherited condition characterized by life threatening heart racing, presenting with palpitations, cardiac arrest (collapse requiring an ambulance) or sudden death. The disease affects the right ventricle, the part of the heart that pumps blood to the lungs. ARVC is diagnosed with a wide range of tests that focus on the pumping function and the electrical signals from the right ventricle. These factors are summarized in a score that forms the ARVC Task Force Criteria. Genetic testing has identified 5 different genes that lead to ARVC, which are detected in about 60% of patients with ARVC. This allows doctors to test family members of the patient with ARVC to determine if they are at risk of developing the condition. Currently, family members undergo testing that includes imaging and electrical tests such as a 24-hour monitor to determine if they have evidence of ARVC. With increasing frequency, family members are found to have the gene that may lead to ARVC, but little or no evidence that their hearts are affected. This may be because the family member is too young to develop the condition, or that other factors that we do not understand have protected them from developing it.

The PREPARE study will study 100 patients that carry a gene that can lead to ARVC, but do not have anything more than minor evidence that the condition is present. These patients will not have heart racing on their initial 24-hour monitor. These patients will undergo long term monitoring with an implanted heart monitor that is inserted with a minor surgical procedure, which will detect abnormal heart rhythms that may provide a clue that heart racing from ARVC is present that is not detected with a 24-hour monitor that is performed on an annual basis (St. Jude Confirm implantable loop recorder). These patients will be enrolled in 10 adult and pediatric centers across Canada, and followed for 3 years after their heart monitor is implanted. If heart racing is detected, patients will discuss these results with their doctor to discuss what it means to them.

DETAILED DESCRIPTION:
Arrhythmogenic Right Ventricular Cardiomyopathy (ARVC) is a familial condition characterized by onset of life threatening ventricular arrhythmias in early adulthood, presenting with ventricular tachycardia, cardiac arrest or sudden death. The disease is diagnosed with tests that focus on imaging the right ventricle and assessing for ambient arrhythmia or abnormal electrical substrate. These factors are collated into a score that forms the ARVC Task Force Criteria, known to be specific but not sensitive. These criteria have been revised in 2010, introducing a broader and more quantitative approach to diagnosis including genetic testing results, intended to enhance sensitivity without reducing specificity. They account for findings from genetic testing, confounded in part by the unknown significance of a positive genetic test in the absence of a phenotype in a disease with variable penetrance and expressivity. Genetic testing identifies the underlying mutation in ≈60% of clearly affected patients. Recent access to genetic testing has demonstrated that family members of an affected individual often harbor the culprit mutation, with little evidence that they are affected from clinical testing. Given the risk of life threatening arrhythmia as a first presentation of disease expression, enhanced detection of ventricular arrhythmia would help to identify patients with manifest ARVC.

The PREPARE study will test the hypothesis that prolonged monitoring with an implantable loop recorder (ILR) will provide evidence of progressive electrical disease in gene positive ARVC patients with a non-diagnostic phenotype (negative or mild) who do not receive an implantable cardioverter defibrillator (ICD). Detection of non-sustained ventricular tachycardia will have incremental value over routine periodic clinical follow-up and standard short term monitoring (24-48 hour Holter).

100 gene positive patients without manifest ARVC after standard screening clinical testing will undergo ILR implantation. These patients will fail to meet 2010 revised Task Force Criteria for definite ARVC and will not be considered candidates for a primary prevention ICD by the local investigator. A Health Canada approved St. Jude Medical ConfirmTM loop recorder will be implanted using standard technique with local anesthetic, and patients will be followed for 3 years. Patients will undergo repeat clinical phenotype testing according to the local institutions standard practice, including testing at 3 years after enrollment to reassess Task Force Criteria (standard care), which will constitute the end of the study. A 24-hour Holter monitor will be encouraged annually to provide standard surveillance for ventricular arrhythmia as a comparator to loop recorder findings. In the event that non-sustained or sustained ventricular tachycardia is detected by the loop recorder (≥8 beats) and/or Holter monitor, clinical assessment by the local investigator will take place to review the tracing and discuss the findings with the patient. This will follow routine clinical care.

The primary end point is detection of ≥8 beats of wide QRS complex tachycardia considered ventricular tachycardia by the ILR. Secondary endpoints will include comparison of ventricular arrhythmia burden between routine surveillance Holter monitoring and the ILR, and change in 2010 Task Force Criteria Score from enrollment to 3-year follow-up.

Patients will provide written informed consent to participate in the study, with data collected in a password-protected web based database. Patients will undergo follow-up at 1 and 4 weeks after implant, at 3 and 6 months and every 6 months thereafter. Follow-up will capture findings from loop recorder interrogation, along with change in clinical status and cardioactive drug use. A 24 Hour Holter monitor will be encouraged annually to provide standard surveillance for ventricular arrhythmia as a comparator to loop recorder findings.

This is a pilot study to explore the prevalence and incidence of ambient asymptomatic ventricular arrhythmias in presymptomatic genotype carriers of ARVC. An empiric number of 100 subjects was chosen based on disease prevalence and recruitment goals. End point adjudication will include a 3 member adjudication committee comprised of coinvestigators. A single interim analysis of end points will be performed by an independent Data and Safety Monitoring Committee after 50 patients have completed at least one year of follow-up.

ELIGIBILITY:
Inclusion Criteria:

1. Identification of a pathogenic mutation† categorized as associated or probably associated with ARVC
2. Failure to meet definite revised Task Force Criteria for ARVC. Mutation carriers by definition have a major criterion, so included patients may have 1 minor criteria, but would meet Task Force Criteria for ARVC with 2 minor criteria or 1 major criterion.
3. < 200 PVCs / hour on screening Holter monitor
4. Age > 2 years

Exclusion Criteria:

1. Implantable device in place (pacemaker, ICD)
2. Age < 2 years
3. Mutation represents a variant of unknown significance with reasonable probability that it may not be disease causing
4. Non-sustained ventricular tachycardia on screening Holter monitor (≥8 beats > 100 bpm) and/or ≥ 200 PVCs / hour
5. Previous syncope or palpitations attributed to ARVC by the site investigator
6. Meets definite revised Task Force Criteria for ARVC (≥2 minor criteria and/or ≥1 additional major criterion). These ARVC patients who do not have an implanted device (ICD or pacemaker) will be included in a parallel voluntary registry separate from the study.

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: ARVC gene carriers with minimal or no evidence of being clinically affected
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2010-12; Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
Detection of ≥8 beats of wide QRS complex tachycardia considered ventricular tachycardia (HR>120 bpm*) by the ILR | 3 year monitoring follow-up
  * an algorithm to determine the ventricular tachycardia detection rate

SECONDARY OUTCOMES:
Comparison of ventricular arrhythmia burden between routine | 3 year monitoring follow-up
  * an algorithm to determine the ventricular tachycardia detection rate
Change in 2010 Task Force Criteria Score from enrollment to 3-year follow-up. | 3 year monitoring follow-up
Detection of ≥30 seconds of wide QRS complex tachycardia considered ventricular tachycardia (HR>120 bpm*). | 3 year monitoring follow-up
Proportion of patients that go on to receive an ICD | 3 year monitoring follow-up
Proportion of patients that develop symptomatic sustained ventricular tachycardia | 3 year monitoring follow-up
Proportion of patients that develop sustained ventricular tachycardia, cardiac arrest or sudden death | 3 year monitoring follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Krahn, MD FRCPC, Principal Investigator — Western University, Canada
Locations (1):
- University of Western Ontario, London, Ontario, Canada